CLINICAL TRIAL: NCT06651255
Title: Algorithm-based Management to Reduce the Recurrence of Gastrointestinal Bleeding and Severe Epistaxis in Von Willebrand Disease: WILL-MANAGE Trial
Brief Title: Algorithm-based Management to Reduce the Recurrence of GI Bleeding and Severe Epistaxis in Von Willebrand Disease
Acronym: WILL-MANAGE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022_0508; 2023-A01508-37 (Other: ANSM)
Record Dates: First submitted 2024-10-18; First posted 2024-10-21 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Von Willebrand Disease (VWD)
Keywords: Von Willebrand disease; gastrointestinal bleeding; angiodysplasia; epistaxis
MeSH Terms: conditions — von Willebrand Diseases; Gastrointestinal Hemorrhage; Angiodysplasia; Epistaxis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Optimized management (Experimental): systematic gastrointestinal and nasal endoscopic exploration, local endoscopic treatment whenever applicable,prophylaxis with stepwise dose escalation of VWF concentrate and use of antiangiogenic drugs in patients with severe GI angiodysplasia-related bleeding
  Interventions: Procedure: Optimized management
- Standard of care management (Other): Standard of care management
  Interventions: Procedure: Standard of care management

INTERVENTIONS:
Procedure: Optimized management — systematic gastrointestinal and nasal endoscopic exploration, local endoscopic treatment whenever applicable,prophylaxis with stepwise dose escalation of VWF concentrate and use of antiangiogenic drugs in patients with severe GI angiodysplasia-related bleeding
  Arms: Optimized management
Procedure: Standard of care management — Standard of care management
  Arms: Standard of care management

SUMMARY:
WILL MANAGE is a prospective multicenter controlled open label randomized trial comparing an algorithm-based multidisciplinary management to a standard of care to reduce the incidence of bleeding (GI bleeding or severe epistaxis) recurrence in von Willebrand disease.

ELIGIBILITY:
Inclusion Criteria:

* Males and females adults aged > 18 years
* With a constitutional von Willebrand Disease (according to the phenotypic criteria of the French Reference Center of von Willebrand Disease)
* With a GI bleeding [either overt (any hematemesis, any melena or hematochezia with at least a 2g/dL drop in hemoglobin) or occult (iron deficiency anemia with at least 2g/dL drop in hemoglobin)] with the presence of angiodysplasia or a negative finding on digestive conventional endoscopy OR with a severe epistaxis (requiring red blood cells transfusion or treatment with VWF concentrates)
* Be affiliated to a social security scheme
* Written informed consent obtained

Exclusion Criteria:

* Acquired von Willebrand Disease
* Presence of an inhibitor to VWF or a contra indication to VWF concentrates
* Contra-indication to videocapsule endoscopy
* Refusal of the procedures part of the study
* Pregnant women or breastfeeding
* Short-life expectancy
* Liver cirrhosis Child-Pugh C or diagnosed portal hypertension
* Cancer currently undergoing chemotherapy
* Inability to provide informed consent
* Patient under justice protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2034-04 (Estimated); Study Completion 2034-12-06 (Estimated)

PRIMARY OUTCOMES:
cumulative incidence of bleeding (GI bleeding or severe epistaxis) recurrence during follow-up | Until the visit 7 (72 months ±2months)
  - GI bleeding is defined as: Any hematemesis or melena Or hematochezia with at least a 2g/dL drop in hemoglobin Or occult bleeding: iron deficiency anemia with at least a 2g/dL drop in hemoglobin
  - Severe epistaxis is defined as: A nose bleed requiring red blood cells transfusion or treatment with VWF concentrates

SECONDARY OUTCOMES:
Number of GI bleeding and severe epistaxis recurrence during follow-up | Until the visit 7 (72 months ±2months)
Number of days of hospitalization for GI bleeding or severe epistaxis recurrence during follow-up | Until the visit 7 (72 months ±2months)
Number of transfused red blood cells units, the total amount of iron supplementation (mg) and number of units of VWF concentrates administred (IU/kg) during follow-up | Until the visit 7 (72 months ±2months)
Change in haemoglobin and serum ferritin levels from inclusion to 3-years | from inclusion to 3-years
Change in bleeding score (ISTH BAT) from inclusion to 3-years. The bleeding score will be calculated for the 3-year period before the evaluation. | from inclusion to 3-years
Change in quality of life assessed by a standardized questionnaire validated for VWD (WISH-QoL scores) from inclusion to 3 years | from inclusion to 3-years

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Susen, MD, Professor, Principal Investigator — Lille University Hospital
Locations (17):
- France (17):
  - CHU Lille, Lille, Nord
  - CHU Tours, Tours, Tours
  - CHU Amiens, Amiens
  - CHRU Brest, Brest
  - Hôpital cardiologique Louis Pradel, Bron
  - CHU Caen, Caen
  - CH Chambery, Chambéry
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CHU Dijon, Dijon
  - AP-HP Hôpital Kremlin Bicetre, Le Kremlin-Bicêtre
  - AP-HM Hôpital Timone, Marseille
  - CHU Montpellier, Montpellier
  - CHU Nantes, Nantes
  - CHU Rennes, Rennes
  - CHU Rouen, Rouen
  - CHU Strasbourg, Strasbourg
  - CHU Toulouse, Toulouse